CLINICAL TRIAL: NCT05537506
Title: Evaluation of Effects of Bracket's Slot System on the Quantity and Quality of Teeth Movements During Orthodontic Leveling and Alignment Stage : A Prospective Clinical Study
Brief Title: Evaluation of Effects of Bracket's Slot System on the Quantity and Quality of Teeth Movements During Orthodontic Leveling and Alignment Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Belal Abdelrahman Abdelmotaleb Elgohary, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 735/1246
Record Dates: First submitted 2022-08-28; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Moderate and Severe Crowding in Lower Dental Arch
Keywords: Slot 0.018; Slot 0.022; Bracket; Leveling; Alignment
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bracket slot 0.018 (Active Comparator)
  Interventions: Device: Bracket slot 0.018
- Bracket slot 0.022 (Active Comparator)
  Interventions: Device: Bracket slot 0.022

INTERVENTIONS:
Device: Bracket slot 0.018 — That includes12 patients who will be treated using the bracket slot 0.018×0.025-inch system.
  Arms: Bracket slot 0.018
Device: Bracket slot 0.022 — Includes12 patients who will be treated using the bracket slot 0.022×0.028-inch system
  Arms: Bracket slot 0.022

SUMMARY:
Evaluation of effect of bracket slot system on the quality and quantity of tooth movement during leveling and alignment stage

ELIGIBILITY:
Inclusion Criteria:

* An age range from14 to18 years. All permanent teeth are erupted(3rd molar not included).
* Angle class I malocclusion with normal facial proportions.
* Moderate to severe crowding in the lower dental arch asassessed by lett irregularity Index that require treatment with fixed appliance using extraction approach.
* There is no previous orthodontic treatment.

Exclusion Criteria:

* Poor oral hygiene or periodontally compromised teeth.
* Craniofacial anomalies or previous history of trauma, bruxism, or Parafunctions.
* Uncooperativepatient.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-08-25 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Rate of tooth movement by different bracket slot system | At 8 months
  Amount of tooth movement

CONTACTS AND LOCATIONS:
Overall Officials: Alazhar University, Principal Investigator — Al-Azhar University
Locations (1):
- Alazhar university, Naşr, Cairo Governorate, Egypt

REFERENCES:
- [Background] Mavragani M, Vergari A, Selliseth NJ, Boe OE, Wisth PL. A radiographic comparison of apical root resorption after orthodontic treatment with a standard edgewise and a straight-wire edgewise technique. Eur J Orthod. 2000 Dec;22(6):665-74. doi: 10.1093/ejo/22.6.665. PMID 11212602